CLINICAL TRIAL: NCT02473991
Title: Correlation Between Placental Thickness in the Second and Third Trimester and Fetal Weight
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, amr elsayed elsayed, researcher for master degree, Ain Shams Maternity Hospital
Other Study IDs: Master degree in Obs & gyn
Record Dates: First submitted 2015-05-10; First posted 2015-06-17 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Pregnancy; Fetal Macrosomia; Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Macrosomia; Fetal Growth Retardation | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — placenta is weighed in grams as described by Azpurua et al.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: ultrasound — The placental thickness was measured by placing the ultrasound transducer perpendicularly to the plane of the placenta, in the area of the cord insertion, near the mid-placental portion

SUMMARY:
The aim of this prospective longitudinal study was to investigate the relationship between placental thickness during the second and third trimesters and placental and birth weights.

DETAILED DESCRIPTION:
The investigator will make certain that the appropriate informed consent process is in place to ensure that potential research subjects, or their authorized representatives, are fully informed about the nature and objectives of the study, the potential risk and benefits of study participation, and their right as research subjects.

All laboratory specimens, evaluation forms, reports, video recordings, and other records that leave the site will not include unique personal data to maintain subject confidentiality.

All patients provided an informed written consent after they were fully instructed about the investigation.The study was approved by ethical committee of Ain Shams University.

All recruited women were observed at the 1st trimester screening at antenatal clinic and assessed for baseline demographic and obstetric data including age, parity, body mass index (BMI) and past medical events. Smoking, alcohol and drug use were also determined.

At second and third trimester (15-20 and 30-34 weeks of gestation respectively), the maternal weight, weight gain, BMI, BMI gain and data of ultrasound examination were recorded. At the time of delivery after assessment of maternal weight as mentioned above, the birth weight (in grams), fetal sex, and mode of delivery were taken.

All pregnant women underwent ultrasound evaluation of placental thickness at the time of second trimester (15-20 weeks of gestation) as well as third trimester (30-34 weeks of gestation).

All sonographic examinations were performed trans-abdominal using a Medison X4 ultrasound machine Trans abdominal4.0 megahertz (MHz) probe at The Special Care Center for Fetus Unit at Ain Shams University Maternity Hospital.

The placental thickness was measured by placing the ultrasound transducer perpendicularly to the plane of the placenta, in the area of the cord insertion, near the mid-placental portion as described by Hoddick et al

Each evaluation was performed by one of two experienced sonographers of our hospital with minimum inter- and intra-observer variability.

After delivery, the placenta was weighed in grams as previously described by Azpurua et al.

Fetal weight (primary objective) and neonatal status and morbidity including baby Apgar scores, fetal distress or fetal death and admission to the neonatal intensive care unit were also determined. All the examinations and data recording were performed by two senior resident physicians.(secondary objective)

ELIGIBILITY:
Inclusion Criteria:

1. patient Aged between 18 and 45 years.
2. singleton viable pregnancy.
3. non scared uterus.

Exclusion Criteria:

1. systemic illness (DM,Hypertension, renal disease, liver disease, sickle cell disease)
2. known congenital fetal anomalies.
3. multiple pregnancy.
4. intra uterine fetal death.
5. anatomical defect of pregnant uterus
6. abnormally located placenta or placental anomalies
7. morbid obesity
8. missing records
9. unwilling to incorporate in the study.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: uncomplicated pregnant women who will attend the outpatient clinic at Ain Shams University Maternity Hospital
Sampling Method: Non-Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AHMED MEKLED, Professor, Study Director — Ain Shams University; HAYTHAM SABAA, Lecturer, Study Director — Ain Shams University
Locations (1):
- Ain shams faculty of medicine, Cairo, Elabbasia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azpurua H, Funai EF, Coraluzzi LM, Doherty LF, Sasson IE, Kliman M, Kliman HJ. Determination of placental weight using two-dimensional sonography and volumetric mathematic modeling. Am J Perinatol. 2010 Feb;27(2):151-5. doi: 10.1055/s-0029-1234034. Epub 2009 Aug 3. PMID 19653142
- [Background] Hoddick WK, Mahony BS, Callen PW, Filly RA. Placental thickness. J Ultrasound Med. 1985 Sep;4(9):479-82. doi: 10.7863/jum.1985.4.9.479. PMID 3903201

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnant Women: All recruited women were observed at the 1st trimester screening at antenatal clinic and assessed for baseline demographic and obstetric data including age, body mass index (BMI).
  All pregnant women underwent ultrasound evaluation of placental thickness at the time of second trimester (15-20 weeks of gestation) as well as third trimester (30-34 weeks of gestation).
  The placental thickness was measured by placing the ultrasound transducer perpendicularly to the plane of the placenta, in the area of the cord insertion, near the mid-placental portion as described by Hoddick et al.(1985).
  At the time of delivery , the birth weight (in grams), and mode of delivery was be taken.
  After delivery, the umbilical cord was immediately clamped at its placental insertion to prevent loss of fetal blood, the maternal surface was dried with a towel, and the membranes were carefully trimmed at the placental margin. Each placenta was weighed within 15 minutes from delivery (Azpurua et al.,2010).
Period: Overall Study
Arm/Group | Pregnant Women
Started | 395
Completed | 395
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pregnant Women
Number analyzed (Participants) | 395
Age, Continuous [Mean (Standard Deviation); unit: years] — the age of participant was between 20 years and 30 years
  years | 25 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 395
  Male | 0
weight [Mean (Standard Deviation); unit: kg] | 78 (12)
Height [Mean (Standard Deviation); unit: Meter] | 1.7 (.07)

OUTCOME MEASURES:

1. Primary Outcome: Fetal Weight (Fetal Weight at Birth)
Description: Fetal weight (fetal weight at birth) (in grams)
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Pregnant Women
Number analyzed (Participants) | 395
gram | 3243 (402)

2. Primary Outcome: Placental Thickness in Second Trimester
Description: placental thickness measured in millimeter
Time Frame: 15-20 weeks of gestation
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Pregnant Women
Number analyzed (Participants) | 395
millimeter | 21.5 (2.5)
Statistical Analysis 1: Comparison: Pregnant Women; Null hypothesis In normal pregnant women, placental thickness during second trimesters may be correlated with birth weight at term; Test type: Superiority or Other; p < 0.01, Regression, Linear

3. Primary Outcome: Placental Thickness at 3rd Trimester
Time Frame: 30-34 weeks of pregnancy
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Pregnant Women
Number analyzed (Participants) | 395
millimeter | 35.6 (4.1)
Statistical Analysis 1: Comparison: Pregnant Women; Null hypothesis In normal pregnant women, placental thickness during third trimesters may be correlated with birth weight at term; Test type: Superiority or Other; p < 0.01, Regression, Linear

ADVERSE EVENTS:
Time Frame: adverse event data collection was about 9 months ( time between starting antenatal care and end delivery )
Arm/Group | Pregnant Women
Serious Adverse Events (participants affected / at risk) | 0/395
Other Adverse Events (participants affected / at risk) | 0/395

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes